CLINICAL TRIAL: NCT02230891
Title: Biomarker Guided Therapies in Stage A/B Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CLNB-009-13F
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Results first posted 2022-09-29 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Hypertension; Diabetes; Cardiovascular Disease
Keywords: heart failure; biomarkers; troponin; BNP; carvedilol; spironolactone; prevention
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Cardiovascular Diseases; Heart Failure | interventions — Carvedilol; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Carvedilol (Active Comparator): Approximately 70 subjects will be randomized to carvedilol
  Interventions: Drug: Carvedilol
- Spironolactone (Active Comparator): Approximately 70 subjects will be randomized to spironolactone
  Interventions: Drug: Spironolactone
- Usual care (Other): Approximately 70 subjects will be randomized to usual care/ standard care by primary care providers
  Interventions: Other: Usual care

INTERVENTIONS:
Drug: Carvedilol — Carvedilol is a non selective beta blocker
  Arms: Carvedilol
Drug: Spironolactone — Spironolactone is an aldosterone antagonist and can lower blood pressure/ is used in heart failure
  Arms: Spironolactone
Other: Usual care — standard care as per primary care provider
  Arms: Usual care

SUMMARY:
Despite advances in cardiovascular care, the occurrence of heart failure (HF) is steadily increasing. The increase in HF rates poses enormous challenges, as once an individual becomes symptomatic or requires hospitalization with HF, the prognosis remains poor. Therefore, prevention of HF is essential. HF prevention is a critical issue as HF risk factors that include common medical conditions such as hypertension and diabetes are also increasing. However, not everyone with these risk factors develops HF. Using novel blood tests, the investigators propose to identify and treat subjects at higher HF risk to see if the investigators can stabilize or improve ultrasound measures known to be associated with HF risk. This study will enroll only Veterans.

DETAILED DESCRIPTION:
Recently the investigators have shown that HF risk prediction can be improved using cardiac troponin T measured with a novel high-sensitivity assay (hs-cTnT) and N-terminal pro-B-type natriuretic peptide (NT-proBNP). Furthermore, hs-cTnT seems to identify individuals at higher risk among those with established risk factors (such as hypertension) for HF. In preliminary results, the investigators have shown that individuals with systolic blood pressure of 120-129 mm Hg and elevated hs-cTnT have a higher rate of incident HF than those with systolic blood pressure of 140-159 mm Hg and undetectable hs-cTnT. Therefore, the investigators believe that by using hs-cTnT to estimate HF risk the investigators can identify individuals in whom aggressive modification of risk factors such as high blood pressure will be associated with a favorable risk-benefit ratio.

The investigators' objective/specific aim therefore is to evaluate if treatment of selected subjects with Stage A or B HF (i.e., those with hs-cTnT >5 ng/L and an estimated 10-year HF hospitalization risk of >5%) who have reasonably well-controlled blood pressure with antihypertensive agents (carvedilol or spironolactone) will be associated with improvement of surrogate markers associated with incident HF (i.e., speckle-tracked cardiac and vascular strain). Carvedilol and spironolactone were chosen for the following reasons: a) they are not routinely used as first-line antihypertensive agents; b) beta-blockade was associated with decreases in hs-cTnT in the preliminary analysis of subjects with established HF; and c) the mechanism of actions of carvedilol and spironolactone provide a sound scientific rationale for use in prevention of HF.

Using a prospective open-label blinded end point (PROBE) design, the investigators propose to randomize 210 subjects aged >40 years with systolic blood pressure between 120-155 mm Hg, cardiac troponin T (measured with a novel high-sensitivity assay) level >5 ng/L, and 10-year HF risk >5% (estimated using a validated laboratory model including demographic factors, NT-proBNP, and hs-cTnT) to receive carvedilol (nonselective beta-blocker), spironolactone (aldosterone antagonist), or usual care for 18 months. The primary end point will be change in global longitudinal systolic myocardial strain estimated using 2D speckle tracking. Additionally, changes in vascular strain and biomarkers will be evaluated. This study will help us identify whether both or either of the medications can be further tested in large randomized clinical trials to prevent the incidence of HF.

ELIGIBILITY:
Inclusion Criteria:

Only Veterans are eligible to participate. Other inclusion criteria include

* Age greater than 40 years
* One of the following in order to establish Stage A HF a. Hypertension b. Diabetes mellitus (controlled: defined as hemoglobin A1c less than 9%) c. Obesity (defined as BMI greater than 30 kg/m2) d. Metabolic syndrome (using the National Cholesterol Education Panel definition) e. Left ventricular hypertrophy (by ECG) f. Coronary or cerebrovascular arterial disease
* Troponin T measured by the high sensitivity assay of greater than 5ng/L
* Systolic BP 120-155 mmHg at primary care provider (PCP) visit and prerandomization visit (i.e., 2 separate confirmations of the same). If there is discordance between the PCP visit and pre-randomization the investigators will bring patient back to recheck his BP and use that as the tie breaker. Not orthostatic with measurements (defined as a fall in systolic BP greater than 20 mmHg when subjects assume an upright position). - Estimated 10-yr HF risk (based on Atherosclerosis Risk in Communities HF Lab model) greater than 5%
* Provides informed consent

Exclusion Criteria:

The exclusion criteria include

* Active Atrial fibrillation
* History of chest/ neck radiation
* High-risk chronic obstructive pulmonary disease (COPD) (GOLD classification 3-4 with greater than equal to 2 COPD exacerbations in the last 12 months)
* Known allergy to carvedilol or spironolactone
* Renal insufficiency with estimated Glomerular Filtration Rate (eGFR) less than 60 ml/min
* Serum potassium greater than 5 meq/L
* Current use of carvedilol, spironolactone, any other beta-blockers or aldosterone antagonists
* Signs of clinical HF on initial examination (pulmonary rales/crackles, elevated jugular venous pulse with S3/S4 on auscultation)
* Left ventricular ejection fraction <50% by echo
* Moderate or greater valve stenosis or regurgitation
* Hypertrophic cardiomyopathy
* Exposure to known cardiotoxic chemotherapy
* Poor echo image quality
* Right ventricular dysfunction more than mild
* Any valvular dysfunction that is more than mild
* Any life-threatening disease expected to result in death within the next 2 years
* Active severe liver disease (evaluated at Visit 1): cirrhosis, active hepatitis, aspartate transaminase (ALT) or alanine transaminase (AST) greater than 3 x ULN, or biliary obstruction with hyperbilirubinemia (total bilirubin greater than 2 x ULN).
* Participation in another clinical trial involving an investigational agent within 90 days prior to randomization
* Any condition or therapy which, in the opinion of the investigator, might pose a risk to the patient or make participation in the study not in the patient s best interest
* Drug or alcohol abuse within the past 6 months, and unable/unwilling to abstain from drug abuse and excessive alcohol consumption during the study. Excessive alcohol consumption is on average greater than 2 units of alcohol per day. A unit of alcohol is defined as a 12-ounce (350 mL) beer, 5-ounce (150 mL) wine, or 1.5-ounce (45 mL) of 80 ]proof alcohol for drinks.
* Mental/psychological impairment or any other reason to expect patient difficulty in complying with the requirements of the study.
* Any immunosuppressed condition where intercurrent illnesses may affect interpretation of study results
* Pregnant women or any woman planning a pregnancy during the study period
* Not meeting any of the inclusion criteria

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Nambi, MBBS, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Carvedilol: Approximately 70 subjects will be randomized to carvedilol
  Carvedilol: Carvedilol is a non selective beta blocker. Dose will be 3.125 mg two times daily with increases in dose if blood pressure permits
- Spironolactone: Approximately 70 subjects will be randomized to spironolactone
  Spironolactone: Spironolactone is an aldosterone antagonist and can lower blood pressure/ is used in heart failure. Spironolactone dose will be 25 mg by mouth once daily
Period: Baseline
Arm/Group | Carvedilol | Spironolactone | Usual Care
Started | 21 | 18 | 19
Completed | 21 | 17 | 18
Not Completed | 0 | 1 | 1
Not completed — Did not meet inclusion | 0 | 1 | 1
Period: 2 Week
Arm/Group | Carvedilol | Spironolactone | Usual Care
Started | 21 | 17 | 0 (No week 2 for subjects in usual care)
Completed | 18 | 15 | 0 (No week 2 for subjects in usual care)
Not Completed | 3 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Consent withdrawn | 1 | 0 | 0
Period: 6 Month
Arm/Group | Carvedilol | Spironolactone | Usual Care
Started | 18 | 15 | 18
Completed | 17 | 12 | 17
Not Completed | 1 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Physician Decision | 0 | 2 | 0
Period: 12 Month
Arm/Group | Carvedilol | Spironolactone | Usual Care
Started | 17 | 12 | 17
Completed | 16 | 9 | 17
Not Completed | 1 | 3 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Period: 18 Month End of Study
Arm/Group | Carvedilol | Spironolactone | Usual Care
Started | 16 | 9 | 17
Completed | 15 | 9 | 16
Not Completed | 1 | 0 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Hear failure, lost to follow up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: These include individuals who participated in the study. Patient who withdrew consent and one who did not meet eligibility criteria and hence was excluded not included
Groups:
- Total: Total of all reporting groups
Arm/Group | Carvedilol | Spironolactone | Usual Care | Total
Number analyzed (Participants) | 20 | 18 | 18 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 3 | 8
  >=65 years | 19 | 14 | 15 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (5.3) | 69.2 (6.5) | 70.6 (5.8) | 70.1 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 20 | 18 | 18 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 9 | 5 | 26
  White | 8 | 9 | 13 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 18 | 58
Baseline troponin [Mean (Standard Deviation); unit: ng/L] — Population: One subject baseline biomarker not available
  ng/L
    number analyzed (Participants) | 19 | 18 | 18 | 55
    (all) | 14.6 (3.3) | 15.4 (4.6) | 17.1 (4.4) | 15.7 (4.2)
N-terminal (NT)-pro hormone BNP (NT-proBNP) [Mean (Standard Deviation); unit: pg/ml] — Population: One subject baseline biomarker not available
  pg/ml
    number analyzed (Participants) | 19 | 18 | 18 | 55
    (all) | 97.0 (78.7) | 72.2 (73.5) | 96.6 (76.4) | 88.7 (75.7)
Pulse wave velocity (PWV) [Mean (Standard Deviation); unit: m/sec] — Population: Based on available data for analysis
  m/sec
    number analyzed (Participants) | 14 | 14 | 13 | 41
    (all) | 10.6 (4.9) | 9.4 (5.5) | 8.5 (4.1) | 9.5 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cardiac Global Longitudinal Strain
Description: Change in myocardial speckle tracked strain (global longitudinal strain) after 18 months (baseline vs. 18 months) of therapy with carvedilol or spironolactone or usual care. The myocardial global longitudinal strain was measured using echocardiography
Time Frame: 18 months
Population: Difference is global longitudinal strain between baseline and 18 months for those who completed both visits and had data available
Measure: Mean (Standard Deviation); unit: % systolic deformation
Arm/Group | Carvedilol | Spironolactone | Usual Care
Number analyzed (Participants) | 15 | 9 | 13
% systolic deformation | -1.4 (4.4) | -1.74 (3.25) | -1.14 (4.13)

2. Secondary Outcome: Change in NTproBNP (Biomarker)
Description: Change in levels of NT-proBNP (measured in blood samples) between baseline and 18 months after therapy with carvedilol or spironolactone or usual care
Time Frame: 18 months
Population: Those who completed study and had data available
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Carvedilol | Spironolactone | Usual Care
Number analyzed (Participants) | 15 | 8 | 14
pg/ml | 87.9 (243.5) | -16.5 (39.3) | 3.65 (91.03)

3. Secondary Outcome: Change in Pulse Wave Velocity
Description: Changes in arterial stiffness between baseline and 18 months after therapy with carvedilol, spironolactone or usual care. Arterial stiffness was measured by pulse wave velocity (Sphygmocor device)
Time Frame: 18 months
Population: Based on available measures at baseline and end of study. Reported values are change in Pulse wave velocity (PWV) between visits
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Carvedilol | Spironolactone | Usual Care
Number analyzed (Participants) | 10 | 8 | 11
m/sec | -0.71 (1.6) | -0.77 (5.7) | -0.59 (3.4)

4. Secondary Outcome: Change in Troponin T Measured Using a High Sensitivity Assay
Description: Change in levels of troponin T (measured with a high sensitivity assay in blood samples) between baseline and 18 months after therapy with carvedilol or spironolactone or usual care
Time Frame: 18 months
Population: Those who completed study and had data available
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Carvedilol | Spironolactone | Usual Care
Number analyzed (Participants) | 15 | 8 | 14
ng/L | -0.2 (5.2) | 1.4 (3.9) | 0.35 (6.0)

ADVERSE EVENTS:
Time Frame: The study had a follow up period of 18 months from randomization during which subjects were followed for adverse events. However, 4 subjects had longer follow up due to the coronavirus infection of 2019 (COVID 19) and inability to schedule follow ups (approximately 6 to 8 months additional follow up for these subjects)
Arm/Group | Carvedilol | Spironolactone | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/21 | 0/18 | 1/19
Serious Adverse Events (participants affected / at risk) | 6/21 | 5/18 | 3/19
Other Adverse Events (participants affected / at risk) | 14/21 | 13/18 | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carvedilol (N=21) | Spironolactone (N=18) | Usual Care (N=19)
Hospitalization for planned surgery (General disorders) | 1 (1) | 1 (2) | 2 (2) — Hospitalizations for planned surgery (hip, cataract, cancer, ablation)
Hospitalization for infection (Infections and infestations) | 0 (0) | 2 (3) | 2 (2) — Infections including pneumonia, COVID, pyelonephritis
Hospitalization for falls, accidents (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) — Falls (mechanical, unclear etc)
Hospitalization for chest pain/ heart failure (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0) — ER visit/ hospitalization for chest pain/ hear failure
Hypotension, ER visit (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) — Low BP needing ER visit
Hospitalization for shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carvedilol (N=21) | Spironolactone (N=18) | Usual Care (N=19)
Breast tenderness (Endocrine disorders) | 0 (0) | 3 (3) | 0 (0)
Renal dysfunction (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (2)
abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Dizziness/ Drowsiness/ Disequilibrium (Cardiac disorders) | 2 (2) | 3 (4) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 6 (10)
chest pain (Cardiac disorders) | 3 (4) | 1 (1) | 1 (2)
Fatigue (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Falls (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Weight loss (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1)
Atrial arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT02230891/Prot_SAP_000.pdf